CLINICAL TRIAL: NCT06066008
Title: Prospective, Dose-Escalating, Investigator Initiated Trial to Evaluate the Safety and Efficacy of ZM-01 in 3-18 Year-old Male Subjects With X-linked Retinoschisis
Brief Title: Safety and Efficacy Study of Novel Gene Therapy ZM-01 for X-linked Retinoschisis Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhongmou Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZM-01
Record Dates: First submitted 2023-09-25; First posted 2023-10-04 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: X-linked Retinoschisis
Keywords: gene therapy; AAV; RS1
MeSH Terms: conditions — Retinoschisis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): IVT administration of a single low dose ZM-01 injection
  Interventions: Drug: ZM-01-L
- group 2 (Experimental): IVT administration of a single high dose ZM-01 injection
  Interventions: Drug: ZM-01-H

INTERVENTIONS:
Drug: ZM-01-L — rAAV-hRS1 intravitreal injection of low dose
  Other Names: rAAV-hRS1
  Arms: group 1
Drug: ZM-01-H — rAAV-hRS1 intravitreal injection of high dose
  Other Names: rAAV-hRS1
  Arms: group 2

SUMMARY:
This trial is meant to evaluate the safety and efficacy of ZM-01 of X-linked retinoschisis. Unilateral intravitreal injections (IVT) will be given into the subject's Study Eye.

DETAILED DESCRIPTION:
X-linked retinoschisis (XLRS) is a rare, inherited retinal disease caused by mutations in the RS1 gene. Individuals affected by XLRS often experience progressive visual impairment from a young age, potentially leading to legal blindness. There is currently no established clinical treatment available. We developed an innovative adeno-associated virus (AAV)-based gene therapy for individuals with XLRS. Six to nine subjects with XLRS received a single unilateral intravitreal injection of ZM-01 at ascending doses.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria will be enrolled into the study

1. Diagnosis of X-linked retinoschisis consistent with the presence of RS1 gene mutation
2. Male, aged between 3 and 18 years old, in overall good health except for XLRS condition
3. Capable of undergoing visual and retinal function assessment.
4. The visual acuity of the study eye not better than: 0.4 (68 ETDRS letters equivalent)
5. No carbonic anhydrase inhibitors have been used at present and for 3 months before treatment
6. Laboratory tests meet the following criteria:

   1. Hemoglobin ≥ 11.0 g/dL
   2. White blood cell counts ranged from 3,300 to 12,000 cells /mm³;
   3. Platelet count 125,000-550,000 /mm³;
   4. Alanine aminotransferase (ALT) is not higher than 1.5 times the upper limit of the normal range of laboratory tests;
   5. Serum creatinine was no higher than 1.1 times the upper limit of the normal range for laboratory tests;
   6. Prothrombin time (PT) ≤14.5 seconds and partial thromboplastin time (PTT) ≤ 36.0 seconds.
7. Willing to discontinue aspirin, aspirin-containing products, and any other medications that may alter clotting function at least 7 days before dosing.
8. Be able to understand and sign informed consent.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria before enrollment were excluded from the study

1. Previously received any AAV gene therapy
2. The following mutations in RS1 gene: R141H, C59S or C223S
3. Pre-existing eye conditions that cause severe vision loss or increase the risk of intravitreal injections (e.g., advanced glaucoma, uveitis, or severe retinal detachment)
4. Ocular diseases in which there is opacity of the lens, cornea, or other media, hindering adequate observation and examination of the retina
5. Use anticoagulant or antiplatelet drugs within 7 days before dosing
6. Use any experimental drug within 3 months prior to registration
7. Presented any situation that causes the investigator to believe the subject might not adhere to the study protocol or that participation might pose an unacceptable risk to the subject

Ages: 3 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2022-09-25 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events | baseline to day 7, month 1, 2
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a product; the event will not need to have a causal relationship with the treatment.
  A serious adverse event (SAE) is any untoward medical occurrence at any dose that leading to the following: Results in death; Life-threatening, refers to an event in which the patient is at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe; Significant or permanent disability/incapacity, where disability refers to a serious disruption and damage of a person's ability to perform normal life functions; Requires inpatient hospitalization or prolongation of existing hospitalization; Congenital anomaly or birth defect; Other medically important events.
Change in best corrected visual acuity (BCVA) | baseline to day 7, month 1, 2
  BCVA of both eyes will be assessed using the early treatment of diabetic retinopathy study (ETDRS) chart or tumbling "E" chart. This approach was chosen to facilitate visual acuity testing in children who cannot recognize letters, which was more appropriate for this study.

SECONDARY OUTCOMES:
Incidence of adverse events and serious adverse events | baseline to month 3, 4, 6, 9, 12
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a product; the event will not need to have a causal relationship with the treatment.
  A serious adverse event (SAE) is any untoward medical occurrence at any dose that leading to the following: Results in death; Life-threatening, refers to an event in which the patient is at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe; Significant or permanent disability/incapacity, where disability refers to a serious disruption and damage of a person's ability to perform normal life functions; Requires inpatient hospitalization or prolongation of existing hospitalization; Congenital anomaly or birth defect; Other medically important events.
Change in Quality of Life | baseline to month 9, 12
  Quality of Life will be measured using Pediatric Eye Questionnaire (PedEyeQ) or other similar questionnaires before and after treatment
Change in best corrected visual acuity (BCVA) | baseline to month 3, 4, 6, 9, 12
  BCVA of both eyes will be assessed using the early treatment of diabetic retinopathy study (ETDRS) chart or tumbling "E" chart. This approach was chosen to facilitate visual acuity testing in children who cannot recognize letters, which was more appropriate for this study.
Change in visual field | baseline to month 1, 2, 3, 4, 6, 9, 12
  Visual field will be assessed by Humphrey perimetry, changes in VFI, MD, PSD will be analyzed.
Change in electrophysiology result | baseline to month 1, 2, 3, 4, 6, 9, 12
  The ERG measurement will be performed based on the standards of international society for clinical electrophysiology of vision (ISCEV).
Anti-AAV neutralizing antibody titer, Anti-RS1 neutralizing antibody titer | baseline to day 1, 7 and month 1, 2
  Peripheral blood samples were collected from each subjects to measure the AAV8 antibody levels and virus titers in the peripheral blood.
Change in the retina cavity assessed by macular OCT | baseline to day 7, month 1, 2, 3, 4, 6, 9, 12
  Optical coherence tomography (OCT) of the macula was performed in both eyes of each participant at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Yin Shen, PhD, Study Chair — Zhongmou Theraputics
Locations (1):
- Wuhan University Renmin Hospital affiliated with Hanchuan Hospital, Xiaogan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
publish research paper